CLINICAL TRIAL: NCT00567944
Title: A Substitute Vestibular Information System Using the BrainPort® Balance Device for Adults With Chronic Vestibular Dysfunction Following Stroke
Brief Title: Use of the BrainPort® Balance Device to Improve Balance in Adults With Balance Deficits Due to Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wicab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCB4-001
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Cerebrovascular Accident
Keywords: Physical Therapy Modalities; Electric Stimulation; Postural Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BrainPort Balance Device — The BrainPort balance device, is a non-invasive medical device that provides head and body position information to a person via their tongue.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the BrainPort balance device in improving balance in people with balance deficits due to stroke.

DETAILED DESCRIPTION:
Following baseline assessments, subjects participate in 5 consecutive days (10 hours) of clinic training with the BrainPort balance device with a Physical Therapist. Assessments are repeated at the end of clinic training. Following clinic training, subjects take the device home to use for two (2) 20 minute training sessions each day. Subjects return to the clinic for one (1) day of testing after using the device at home for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Diagnosis of stroke for at least 6 months.
* Reached a plateau and been discharged from physical therapy.
* Able to ambulate with or without assistance.
* Ongoing balance problem.
* Able to read and understand the informed consent form, and willing to sign the informed consent form.

Exclusion Criteria:

* Current oral health problems as determined by health questionnaire and an examination of the oral cavity.
* Any medical condition that would interfere with performance on the assessments.
* History of seizures.
* Pregnancy.
* Cognitive deficits (Mini-Mental 25 or below), joint replacements, cervical vertigo, or major neurologic disease, major depression or disabling psychiatric disorder.
* Known neuropathies of tongue or skin tactile system.
* Prior exposure to BrainPort® balance device.
* Subjects who are unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests, and return to clinic for a follow-up visit.
* Subjects who have undergone middle ear or other surgery with sacrifice or damage to the chorda tympani nerve, lingual nerve, or hypoglossal nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | baseline, 5 days, end of study
Berg Balance Scale | Baseline, 5 days, end of study
Activities-specific Balance Confidence Scale | Baseline, 5 days, end of study
Timed Up and Go | Baseline, 5 days, end of study
Stroke Impact Scale | Baseline, 5 day, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Badke, PT, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Middleton, Wisconsin, United States

REFERENCES:
- [Background] Bach-y-Rita P, W Kercel S. Sensory substitution and the human-machine interface. Trends Cogn Sci. 2003 Dec;7(12):541-6. doi: 10.1016/j.tics.2003.10.013. PMID 14643370
- [Background] Bach-Y-Rita P. Emerging concepts of brain function. J Integr Neurosci. 2005 Jun;4(2):183-205. doi: 10.1142/s0219635205000768. PMID 15988797
- [Background] Tyler M, Danilov Y, Bach-Y-Rita P. Closing an open-loop control system: vestibular substitution through the tongue. J Integr Neurosci. 2003 Dec;2(2):159-64. doi: 10.1142/s0219635203000263. PMID 15011268
- [Background] Danilov Y, Tyler M. Brainport: an alternative input to the brain. J Integr Neurosci. 2005 Dec;4(4):537-50. doi: 10.1142/s0219635205000914. PMID 16385646
- See also: Wicab Inc. homepage — http://www.wicab.com